CLINICAL TRIAL: NCT04664972
Title: Comparing TP (Docetaxel + Cisplatin) and TAC (Docetaxel + Doxorubicin + Cyclophosphamide) in Neoadjuvant Therapy for Operable Triple Negative Breast Cancer, A Multicenter, Randomized, Phase II Clinical Trial
Brief Title: Comparison of TP and TAC Regimens in Neoadjuvant Treatment of TNBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Director, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HELEN-001
Record Dates: First submitted 2020-11-09; First posted 2020-12-11 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAC regimen group (Placebo Comparator): The control group was treated with TAC (docetaxel 75mg/m2 + adriamycin 50mg /m2 + cyclophosphamide 500mg/m2) for 6 cycles, 21 days as a cycle.
  Interventions: Drug: Docetaxel +doxorubicin+ cyclophosphamide
- TP regimen group (Experimental): The experimental group was treated with TP (docetaxel 75mg/m2 day 1 + cisplatin 25 mg/m2 day 1,2,3) neoadjuvant chemotherapy for 6 cycles, 21 days as a cycle.
  Interventions: Drug: Docetaxel +Cisplatin

INTERVENTIONS:
Drug: Docetaxel +doxorubicin+ cyclophosphamide — The control group was treated with TAC (docetaxel 75 mg / m2 + adriamycin 50 mg / m2 + cyclophosphamide 500 mg / m2) for 6 cycles, 21 days was a cycle.
  Other Names: TAC regimen group
  Arms: TAC regimen group
Drug: Docetaxel +Cisplatin — The experimental group was treated with TP (docetaxel 75mg/m2 day 1 + cisplatin 25 mg/m2 day 1,2,3) neoadjuvant chemotherapy for 6 cycles, 21 days as a cycle.
  Other Names: TP regimen group
  Arms: TP regimen group

SUMMARY:
Previous studies have shown that TNBC is sensitive to DNA crosslinking-related chemotherapeutic drugs such as platinum. However, there is a lack of large sample prospective clinical data to compare the efficacy of TP and EC-T / TEC regimen in the neoadjuvant chemotherapy of TNBC. Besides, the application of anthracycline drugs is limited to a certain extent due to the cardiotoxicity. Based on the above evidence, the researchers hope to explore a more effective and safer new adjuvant therapy for TNBC.

DETAILED DESCRIPTION:
In this study, TNBC patients were randomly divided into experimental group and control group, the ratio of experimental group to control group was 1:1. The experimental group received 6 cycles of neoadjuvant chemotherapy (docetaxel 75 mg / m2 day 1 + cisplatin 25 mg / m2 day 1, 2, 3), 21 days as a cycle. The control group was treated with TAC (docetaxel 75mg / M2 + adriamycin 50mg / M2 + cyclophosphamide 500mg / m2) for 6 cycles, 21 days as a cycle. To compare the efficacy and safety of 6*TP (docetaxel + cisplatin) regimen and traditional 6*TAC (docetaxel + doxorubicin + cyclophosphamide) regimen in neoadjuvant chemotherapy of TNBC.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70.
2. Clinical stage Ⅱ-Ⅲ.
3. triple negative and invasive breast cancer confirmed by histopathology:

   Triple negative breast cancer is defined as:
   * negative for ER and PR (IHC nuclear staining < 10%).
   * Her-2 negative (IHC 0,1 + without FISH, or IHC 2 + and without FISH amplification).
4. With clinically measurable focus: Measurable lesions observed on ultrasound, mammography, or magnetic resonance imaging (optional) within the month prior to randomization.
5. Organ and bone marrow function tests within 1 month before chemotherapy indicate no contraindications to chemotherapy:

   * neutrophils count absolute value ≥ 2.0×109/L
   * hemoglobin ≥ 100g/L
   * blood platelet ≥ 100×109/L
   * total bilirubin < 1.5 ULN (upline of normal value)
   * creatinine < 1.5×ULN
   * AST/ALT < 1.5×ULN;
6. Cardiac ultrasound EF value ≥ 55%.
7. Females of childbearing age with negative serum pregnancy test 14 days before randomization.
8. ECOG score ≤1.
9. Sign informed consent.

Exclusion Criteria:

1. Evidence of metastatic breast cancer (excluding metastatic breast cancer, a chest CT, abdominal ultrasound, or CT and bone scanning should be performed at any time point before diagnosis and randomization; PET/CT scanning can be used as an alternative imaging examination mean) .
2. The patients have received chemotherapy, endocrine therapy, targeted therapy, and radiation therapy for this disease.
3. The patient has a second primary malignant tumor, except for:

   - Thoroughly treated skin cancer
4. Due to severe and uncontrollable other medical diseases, researchers believe the existence of chemotherapy contraindications.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2022-11-26 (Actual); Study Completion 2022-11-26 (Actual)

PRIMARY OUTCOMES:
The pathological complete remission rate (pCR rate) | Immediately after surgery
  Pathological complete response rate (PCR rate), which means there is no invasive cancer (i.e. ypT0/is, ypN0) in the excised specimen (breast+lymphnode) following neoadjuvant chemotherapy and surgery.

SECONDARY OUTCOMES:
Event free survival rate (EFS) | 5 years after surgery
  Time from randomization to any of the following events: disease progression during neoadjuvant therapy, local or remote recurrence, second primary malignant tumor (breast cancer or other cancers) or death from any cause.
Clinical response rate (CRR) | before breast cancer surgery
  CRR judged based on RECIST v1.1
Breast -conserving rate | up to 24 weeks
  Breast -conserving rate
Number of adverse events and serious adverse events | After each cycle of chemotherapy (21 days as 1 cycle)
  Evaluate the nature, incidence and severity of chemotherapy adverse events according to CTCAE 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhen Liu, Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China